CLINICAL TRIAL: NCT05334160
Title: Evaluation of the Postoperative Effects of Preoperative Abdominal Breathing Exercises in Laparoscopic Cholecystectomy Operations
Brief Title: Pain and Abdominal Breathing Exercises
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, M.D, Tokat Gaziosmanpasa University
Other Study IDs: 21-KAEK-230
Record Dates: First submitted 2022-04-10; First posted 2022-04-19 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Analgesia; Breathing
MeSH Terms: conditions — Agnosia; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative evaluation of patients who did and did not do preoperative abdominal breathing exercises.

DETAILED DESCRIPTION:
The respiratory type and pattern of all patients will be recorded before gallbladder surgery.

In Group P, abdominal breathing training will be given to the patients in this group. They will perform abdominal breathing for at least 5 minutes 6 times a day until surgery.

In Group C,patients who are not given abdominal breathing.

In the intraoperative period, 10 mg / kg paracetamol and 0.05 mg / kg morphine will be used for postoperative analgesia. After surgery, all patients will be given 10 mg/kg paracetamol every 8 hours and will be fitted with a patient-controlled analgesia (PCA) device (Tramadol HCL). PCA device bolus dose will be set to 20 mg, lock time will be set to 10 minutes and the number of buttons per hour will be set as 3.for postoperative analgesia.After surgery, NRS scores of the patients will be evaluated (in the recovery room, 1,2,6,12 and 24 hours.

Preoperative anxiety, postoperative discharge time and analgesic consumption of all patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Planned to gall bladder surgery
* An American Society of Anesthesiologists score of 1,2 or 3

Exclusion Criteria:

* Severe cardiovascular disease
* Respiratory disease
* Psychiatric disease
* Those who have chronic pain

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gallbladder surgerysurgery patients who will be operated under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | During postoperative up to 24 hours
NRS | During postoperative up to 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Hakan Tapar, Tokat Province, Turkey (Türkiye)